CLINICAL TRIAL: NCT02294318
Title: HealthCall: Brief Intervention to Reduce Drug Use in HIV Primary Care
Brief Title: HealthCall-S: A Pilot Study Targeting Concurrent Non-injection Drug Use and Alcohol in HIV Primary Care Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Responsible Party: Principal Investigator, Efrat Aharonovich, Research Scientist V, Research Foundation for Mental Hygiene, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA024606-S
Record Dates: First submitted 2014-11-17; First posted 2014-11-19 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Alcohol or Other Drugs Use
MeSH Terms: conditions — Substance-Related Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motivational Interviewing (MI) (Active Comparator): Participants will engage in a 30-minute Motivational Interviewing session with the study counselor to discuss participant's drug and alcohol use, its implications for their health, and the possibility of drug and alcohol use reduction. This counseling session is intended to help people reduce their drug and alcohol use if they wish. In the counseling session, participants describe the pros and cons of their drug and alcohol use and whether it might be important to quit using drugs and drinking alcohol. Open discussion of the pros (what they like about drug use and drinking) and cons (what they don't like) can help people think about reducing drug and alcohol use in a more complete way than they might have before. This arm will be compared to the HealthCall+Motivational Interviewing arm.
  Interventions: Behavioral: Motivational Interviewing
- HealthCall+Motivational Interviewing (Experimental): The HealthCall+Motivational Interviewing arm will investigate whether the addition of HealthCall, a smartphone application designed to keep track of the participant's drug and alcohol use and other health-related behaviors through short daily use, will help participants reduce their substance use more than Motivational Interviewing alone. Participants will receive the same 30-minute Motivational Interviewing session as described in the MI arm. After the session, participants will be introduced to HealthCall and will be asked to use the app daily over the next 30 days. Each use lasts 2-3 minutes and can be done anywhere on the phone in the U.S. The purpose of daily HealthCall use is to help participants keep track of their drug and alcohol use.
  Interventions: Behavioral: HealthCall+Motivational Interviewing

INTERVENTIONS:
Behavioral: HealthCall+Motivational Interviewing — HealthCall is a technology-based enhancement to brief MI to improve behavior outcomes. It is introduced to patients by the study counselor at the end of the MI session.
  Other Names: MI+HealthCall
  Arms: HealthCall+Motivational Interviewing
Behavioral: Motivational Interviewing — Motivational Interviewing is a client-centered counseling approach for eliciting behavior change.
  Arms: Motivational Interviewing (MI)

SUMMARY:
This pilot study goal is to compare two different treatments to help HIV positive patients reduce their concurrent drinking and non-injection drug use.

DETAILED DESCRIPTION:
The goal of this study is to compare the effects of brief motivational interviewing with participation in HealthCall to brief motivational interviewing alone on non-injection drug and alcohol use. HealthCall involves 2-3 minutes of daily smartphone use to track drug use, drinking behaviors and other aspects of health, followed by personalized feedback in a graph after 30 and 60 days of using the smartphone.

ELIGIBILITY:
Inclusion Criteria:

Age 18 and older; 2. During the prior 30 days, > 4 days of non-injection of cocaine, methamphetamine or heroin, one of which is identified by the patient as his/her primary drug During prior 30 days, > 1 day of binge drinking (>4 drinks on one occasion); Completion of medically supervised detoxification if such detoxification is required; HIV Positive ; Able to give informed consent

Exclusion Criteria:

Patient is currently psychotic, suicidal, or homicidal. Patient has injected any drug in the last 6 months Patient has definite plans to leave the greater New York metropolitan area within the study period.

Patient has gross cognitive/psychomotor impairment as evidenced on the Halstead-Reitan Trails (A+B) Patient does not speak English or Spanish Patient has a hearing and/or vision impairment that precludes smartphone use.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Efrat Aharonovich, PhD, Principal Investigator — The New York State Psychiatric Institute
Locations (1):
- The New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Background] Hasin DS, Aharonovich E, O'Leary A, Greenstein E, Pavlicova M, Arunajadai S, Waxman R, Wainberg M, Helzer J, Johnston B. Reducing heavy drinking in HIV primary care: a randomized trial of brief intervention, with and without technological enhancement. Addiction. 2013 Jul;108(7):1230-40. doi: 10.1111/add.12127. Epub 2013 Apr 17. PMID 23432593
- [Background] Aharonovich E, Greenstein E, O'Leary A, Johnston B, Seol SG, Hasin DS. HealthCall: technology-based extension of motivational interviewing to reduce non-injection drug use in HIV primary care patients - a pilot study. AIDS Care. 2012;24(12):1461-9. doi: 10.1080/09540121.2012.663882. Epub 2012 Mar 20. PMID 22428809
- [Result] Aharonovich E, Stohl M, Cannizzaro D, Hasin D. HealthCall delivered via smartphone to reduce co-occurring drug and alcohol use in HIV-infected adults: A randomized pilot trial. J Subst Abuse Treat. 2017 Dec;83:15-26. doi: 10.1016/j.jsat.2017.09.013. Epub 2017 Sep 29. PMID 29129192

RESULTS

PARTICIPANT FLOW:
Groups:
- HealthCall+Motivational Interviewing: The HealthCall+Motivational Interviewing arm will investigate whether the addition of HealthCall, a smartphone application designed to keep track of the participant's drug and alcohol use and other health-related behaviors through short daily use, will help participants reduce their substance use more than Motivational Interviewing alone. Participants will receive the same 30-minute Motivational Interviewing session as described in the MI arm. After the session, participants will be introduced to HealthCall and will be asked to use the app daily over the next 30 days. Each use lasts 2-3 minutes and can be done anywhere on the phone in the U.S. The purpose of daily HealthCall use is to help participants keep track of their drug and alcohol use.
  HealthCall+Motivational Interviewing (MI): HealthCall is a technology-based enhancement to brief MI to improve behavior outcomes. It is introduced to patients by the study counselor at the end of the MI session.
Period: Overall Study
Arm/Group | Motivational Interviewing (MI) | HealthCall+Motivational Interviewing
Started | 24 | 23
Completed | 21 | 21
Not Completed | 3 | 2
Not completed — Worsening of drinking | 3 | 0
Not completed — Not exposed to intervention | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motivational Interviewing (MI) | HealthCall+Motivational Interviewing | Total
Number analyzed (Participants) | 24 | 23 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.92 (7.21) | 51 (7.02) | 50.96 (7.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 19 | 17 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 21 | 18 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 18 | 37
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 23 | 47

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Days Used Primary Drug (NumDU)
Description: This outcome was derived from a Timeline Follow Back (TLFB) completed at the end of the intervention (day 60).
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Motivational Interviewing (MI) | HealthCall+Motivational Interviewing
Number analyzed (Participants) | 21 | 23
days | 8.5 (6.1) | 5.0 (5.7)

2. Primary Outcome: Mean Dollar Amount Spent Per Day on Primary Drug (QuantU)
Description: This outcome was derived from a Timeline Follow Back (TLFB) completed at the end of the intervention (day 60).
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Motivational Interviewing (MI) | HealthCall+Motivational Interviewing
Number analyzed (Participants) | 21 | 23
dollars | 14.6 (12.7) | 7.1 (9.0)

3. Primary Outcome: Mean Number of Drinking Days (NumDD)
Description: This outcome was derived from a Timeline Follow Back (TLFB) completed at the end of the intervention (day 60).
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Motivational Interviewing (MI) | HealthCall+Motivational Interviewing
Number analyzed (Participants) | 21 | 23
days | 8.1 (5.7) | 7.0 (7.6)

4. Primary Outcome: Mean Number of Drinks Per Day (QuantDD)
Description: This outcome was derived from a Timeline Follow Back (TLFB) completed at the end of the intervention (day 60).
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: standard drinks
Arm/Group | Motivational Interviewing (MI) | HealthCall+Motivational Interviewing
Number analyzed (Participants) | 21 | 23
standard drinks | 1.3 (1.1) | .9 (1)

ADVERSE EVENTS:
Time Frame: through study completion, an average of 60 days
Arm/Group | Motivational Interviewing (MI) | HealthCall+Motivational Interviewing
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 3/24 | 0/23
Other Adverse Events (participants affected / at risk) | 0/24 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Motivational Interviewing (MI) (N=24) | HealthCall+Motivational Interviewing (N=23)
worsening of alcohol use (Psychiatric disorders) | 3 (3) | 0 (0) — Three participants assigned to MI-only entered inpatient alcohol detoxification immediately after randomization due to acute worsening of their drinking.

LIMITATIONS AND CAVEATS:
Recruitment limited to an outpatient clinic in urban setting only. Study does not provide information about patients presenting with severe withdrawal who might benefit from HealthCall once condition is resolved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No